CLINICAL TRIAL: NCT04716972
Title: Evaluating the Impact of COVID-19 on Research in Care Homes
Brief Title: Evaluating the Impact of COVID-19 (Coronavirus) on Research in Care Homes
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021COV114
Record Dates: First submitted 2021-01-18; First posted 2021-01-20 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Online Survey: Online survey
  Interventions: Other: survey
- Interviews: Interviews
  Interventions: Other: Interview

INTERVENTIONS:
Other: survey — Online survey
  Groups: Online Survey
Other: Interview — Interview
  Groups: Interviews

SUMMARY:
During the COVID-19 (corona virus) pandemic the research arena has had to rapidly adapt and change in order to facilitate and deliver research. The UK (United Kingdom) government and Public Health England have stressed the importance of such research to find solutions to treating, preventing and stopping the spread of COVID-19. Due to national and international 'lock down restrictions' delivering research in care home settings has become even more challenging. The adaptations to conducting consultations have relied heavily on the use of technology, for example video calling, telephone, email, and teleconferencing. It is suggested that the use of technology in care home settings is already a barrier to effective research delivery.

Nevertheless, as care home residents are a vulnerable group, it is critical to include these groups in research in order to enable improved and evidence-based care and their access to new and emerging treatments.

This study aims to assess the opinions and experiences of key stakeholders to identify barriers, and enable better facilitation of research in these settings during and post pandemic.

DETAILED DESCRIPTION:
This two phase project will use a mixed methodology.

Phase one will involve mixed methods surveys. One will be completed by care home residents and the other will be completed by research delivery staff and care home staff.

Phase two will involve qualitative interviews with each of these groups to enable better insight into their views and opinions on research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Any resident of a care home in the West Midlands
* Any relative/friend of a care home resident in the West Midlands
* Any staff member or volunteer working in care home in the West Midlands
* Any researcher undertaking research in a care home in the West Midlands (during the pandemic or proposed during the pandemic period)

Exclusion Criteria:

* Individuals who are unable to give Informed Consent
* Individuals who lack capacity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any staff member working/volunteering in a care home, research staff, residents of care homes, relatives of care home residents, all across the West Midlands are eligible to take part in this research project.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of vaccine studies in the care home setting through feedback questionnaire with loose themes and no unique measurements. | 6 months
  To inform the design and delivery of vaccine studies in the care home setting, ensuring they are acceptable by key stakeholders
Acceptability of vaccine studies in the care home setting through feedback interview with loose themes and no unique measurements | 6 months
  To inform the design and delivery of vaccine studies in the care home setting, ensuring they are acceptable by key stakeholders
Acceptability of new ways of delivering research through explorative interview with loose themes and no unique measurements | 6 months
  To inform and assess the acceptability of new ways of delivering research in care home settings, guiding changes and implementation of new ways of working moving forward
Acceptability of new ways of delivering research through explorative questionnaire with loose themes and no unique measurements | 6 months
  To inform and assess the acceptability of new ways of delivering research in care home settings, guiding changes and implementation of new ways of working moving forward

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hard, Principal Investigator — National Institute for Health Research, United Kingdom
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No